CLINICAL TRIAL: NCT04771286
Title: A Phase I, Open-label, Non-randomized, Single-dose, Single-arm, Single-period Study to Investigate the Metabolism and Pharmacokinetics of [C-14]-Labelled BI 1015550 After Oral Administration in Healthy Male Subjects
Brief Title: A Study in Healthy Men to Find Out How BI 1015550 is Taken up and Handled by the Body
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1305-0016; 2020-005934-13 (EudraCT Number)
Record Dates: First submitted 2021-02-23; First posted 2021-02-25 (Actual); Results first posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-10

CONDITIONS: Healthy
MeSH Terms: interventions — BI 1015550; Carbon-14

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BI 1015550 (C-14) (Experimental): Participants received a single dose of 18 milligrams (mg) BI 1015550 (C-14) consisting of 17.16 mg non-labelled BI 1015550 mixed with 0.84 mg [14C]BI 1015550-EQ as 36 milliliters (mL) of oral solution (0.5 mg/mL) labelled with a radioactive dose of 3.7 megaBecquerel (MBq) (100 micro Curie (μ Ci), corresponding to 0.2864 miliSievert (mSV)) on Day 1 with 240 mL of water after an overnight fast of at least 10 hours.
  Interventions: Drug: BI 1015550 (C-14)

INTERVENTIONS:
Drug: BI 1015550 (C-14) — BI 1015550 (C-14)
  Other Names: Nerandomilast; JASCAYD®

SUMMARY:
The main objective of this trial is to investigate the basic pharmacokinetics of BI 1015550 and its metabolite BI 764333 (M480), [14C]-radioactivity, including mass balance, excretion pathways and metabolism following a single oral dose BI 1015550 (C-14) administered to healthy male subjects.

The primary objective is:

- To assess the mass balance recovery of [14C]-radioactivity from urine and faeces as well as vomit in case of occurrence after a single oral dose of BI 1015550 (C-14) administered to healthy male subjects

The secondary objectives are:

* To assess the pharmacokinetics of [C-14]-BI 1015550 and BI 1015550 as well as its metabolite BI 764333 in plasma following a single oral dose of BI 1015550 (C-14)
* To assess the safety and tolerability of BI 1015550

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiograms (ECG), and clinical laboratory tests
* Age of 18 to 65 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent prior to admission to the study, in accordance with Good Clinical Practice (GCP) and local legislation
* Male subjects who meet any of the following criteria from screening until 90 days after trial completion:

  * Use of adequate contraception of the female partner, e.g. any of the following methods plus condom: implants, injectables, combined oral or vaginal contraceptives, intrauterine device, which started at least two months prior to first study drug administration or barrier method (e.g. diaphragm with spermicide) or,
  * Sexually abstinent or,
  * A vasectomy performed at least 1 year prior to screening (with medical assessment of the surgical success) or,
  * Surgically sterilised female partner (including hysterectomy, bilateral tubal occlusion, or bilateral oophorectomy) or,
  * Postmenopausal female partner, defined as at least 1 year of spontaneous amenorrhea (in questionable cases a blood sample with levels of Follicle-Stimulating Hormone (FSH) above 40 U/L and estradiol below 30 ng/L is confirmatory)

Exclusion Criteria:

* Any finding in the medical examination (including blood pressure (BP), pulse rate (PR) or electrocardiogram (ECG)) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 millimetre of mercury (mmHg), diastolic blood pressure outside the range of 45 to 90 mmHg, or pulse rate outside the range of 40 to 100 (beats per minute) bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Further exclusion criteria apply

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2021-05-17 (Actual); Study Completion 2021-05-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- ICON, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a phase I, open-label, non-randomized, single-dose, single-arm, single-period study to investigate the basic pharmacokinetics (PK) of BI 1015550 and its metabolite BI 764333 (M480), [14C]-radioactivity, including mass balance, excretion pathways, and metabolism following a single oral dose of BI 1015550 (C-14) administered to healthy male subjects.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- BI 1015550 (C-14): Participants received a single dose of 18 milligram (mg) BI 1015550 (C-14) consisting of 17.16 mg non-labelled BI 1015550 mixed with 0.84 mg [14C]BI 1015550-EQ as 36 milliliters (mL) of oral solution (0.5 mg/mL) labelled with a radioactive dose of 3.7 megaBecquerel (MBq) (100 micro Curie (μ Ci), corresponding to 0.2864 miliSievert (mSV)) on Day 1 with 240 mL of water after an overnight fast of at least 10 hours.
Period: Overall Study
Arm/Group | BI 1015550 (C-14)
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The TS set included all subjects who were entered and treated with the single dose of the trial drug.
Arm/Group | BI 1015550 (C-14)
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.3 (17.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of the Amount of [14C]-Radioactivity Excreted Among the Administered Single Oral Dose of [14-C] BI 1015550-EQ in Urine (Feurine, 0-tz), Faeces (Fefaeces, 0-tz) and Vomit (Fevomit, 0-tz)
Description: 0-tz refers to 0 until latest individually available cumulative fraction after drug administration.
  Vomit=Not applicable. Amount excreted calculated by volume multiplied with concentration of sample for respective time interval. Amount then refers to administered dose as fraction excreted in percent (dose=100%), done cumulatively.
  Time frames:
  Urine: on Day -1 or 1 -2 hours (h) before drug administration + at 0-4, 4-8, 8-12, 12-24, 24-48, 48-72, 72-96, 96-120, 120-144, 144-168, 168-192, 192-216 h after drug administration.
  Faeces: on Day -1 or 1 -2 hours (h) before drug administration + 0-24, 24-48, 48-72, 72-96, 96-120, 120-144, 144-168, 168-192, 192-216 h after drug administration.
  Thereafter, if warranted, 24 h collections for urine and faeces were to be performed every 7 days starting on Day 16, at Day 16-17, Day 23-24, Day 30-31. When the release criteria for radioactivity recovery had been met then urine/faeces sampling was stopped (earliest stop on Day 10).
Time Frame: From Day -1 or Day 1 - 2 hours (h) before drug administration until release criteria for radioactivity recovery had been met, up to Day 30-31. See also description section.
Population: Treated set (TS): The TS set included all subjects who were entered and treated with the single dose of the trial drug. There was no occurrence of vomit among the participants therefore number of participants analyzed is zero for fevomit,0-tz.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of administered dose
Arm/Group | BI 1015550 (C-14)
Number analyzed (Participants) | 6
Percentage of administered dose
  urine | 36.4 (11.8)
  faeces | 58.0 (12.7)
  vomit: number analyzed (Participants) | 0

2. Secondary Outcome: Area Under the Concentration-time Curve of BI 1015550 in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of BI 1015550 in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) is presented.
Time Frame: Within 2 hours (h) before drug administration and 30 minutes (min), 45 min, 1h, 1h 30 min, 2h, 4h, 8h, 12h, 24h, 36h, 48h, 96h, 144h, 168h, 192h and 216h after drug administration.
Population: Pharmacokinetic parameter analysis set (PKS): PKS included all subjects in TS who provided at least 1 pharmacokinetics (PK) endpoint that was defined as primary or secondary and was not excluded due to protocol violation relevant to evaluation of PK or due to PK non-evaluability. Thus, a subject was included in the PKS, even if the subject contributed only 1 PK parameter value for 1 period to the statistical assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanomole/Liter
Arm/Group | BI 1015550 (C-14)
Number analyzed (Participants) | 6
hours*nanomole/Liter | 2850 (19.5)

3. Secondary Outcome: Area Under the Concentration-time Curve of BI 764333 in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of BI 764333 in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) is presented.
  BI 764333 is a metabolite of BI 1015550.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanomole/Liter
Arm/Group | BI 1015550 (C-14)
Number analyzed (Participants) | 6
hours*nanomole/Liter | 672 (32.9)

4. Secondary Outcome: Area Under the Concentration-time Curve of [14-C] BI 1015550-EQ in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of [14-C] BI 1015550-EQ in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) is presented.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanomole/Liter
Arm/Group | BI 1015550 (C-14)
Number analyzed (Participants) | 6
hours*nanomole/Liter | 10600 (25.6)

5. Secondary Outcome: Maximum Measured Concentration of BI 1015550 in Plasma (Cmax)
Description: Maximum measured concentration of BI 1015550 in plasma (Cmax) is presented.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole/Liter
Arm/Group | BI 1015550 (C-14)
Number analyzed (Participants) | 6
nanomole/Liter | 544 (11.8)

6. Secondary Outcome: Maximum Measured Concentration of BI 764333 in Plasma (Cmax)
Description: Maximum measured concentration of BI 764333 in plasma (Cmax) is presented. BI 764333 is a metabolite of BI 1015550.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole/Liter
Arm/Group | BI 1015550 (C-14)
Number analyzed (Participants) | 6
nanomole/Liter | 13.0 (29.2)

7. Secondary Outcome: Maximum Measured Concentration of [14-C] BI 1015550-EQ in Plasma (Cmax)
Description: Maximum measured concentration of [14-C] BI 1015550-EQ in plasma (Cmax) is presented.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole/Liter
Arm/Group | BI 1015550 (C-14)
Number analyzed (Participants) | 6
nanomole/Liter | 606 (12.4)

8. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAE)
Description: Percentage of participants with treatment-emergent adverse events (TEAE) is presented.
  Percentages were rounded to one decimal place.
Time Frame: From the first administration of the trial drug until end of the trial, up to 31 days.
Population: Treated set (TS): The TS set included all subjects who were entered and treated with the single dose of the trial drug.
Measure: Number; unit: Percentage of participants
Arm/Group | BI 1015550 (C-14)
Number analyzed (Participants) | 6
Percentage of participants | 66.7

ADVERSE EVENTS:
Time Frame: "All-Cause Mortality", "Serious Adverse Events", and "Other Adverse Events": From the first administration of the trial drug until end of the trial, up to 31 days.
Description: Treated set (TS): The TS set included all subjects who were entered and treated with the single dose of the trial drug.
Arm/Group | BI 1015550 (C-14)
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 4/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 1015550 (C-14) (N=6)
Abdominal discomfort (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Headache (Nervous system disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-01-28): https://cdn.clinicaltrials.gov/large-docs/86/NCT04771286/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-29): https://cdn.clinicaltrials.gov/large-docs/86/NCT04771286/SAP_001.pdf